CLINICAL TRIAL: NCT03097198
Title: Effect of Plum-blossom Needle vs. Tropicamide Eye Drops on Juvenile Myopia: A Cross-over Single-blind Randomized Study
Brief Title: Effect of Plum-blossom Needle vs. Tropicamide Eye Drops on Juvenile Myopia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Tang Lewei, Principal Investigator, Wenzhou Medical University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2016ZB080
Record Dates: First submitted 2017-03-20; First posted 2017-03-31 (Actual); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Myopia
Keywords: Juvenile; Traditional Chinese Medicine; Plum-blossom needle
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PbN-TED (Experimental): Treated with plum-blossom needle first for 10 times during 20 days, followed with a one-month wash-out period and a 10-day period with Tropicamide Eye Drops.
  Interventions: Other: Plum-blossom Needle; Drug: Tropicamide Eye Drops
- TED-PbN (Experimental): Treated with Tropicamide Eye Drops for 10 days first, followed with a one-month wash-out period and 10 times of plum-blossom needle treatment for 20 days.
  Interventions: Other: Plum-blossom Needle; Drug: Tropicamide Eye Drops

INTERVENTIONS:
Other: Plum-blossom Needle — * acupoint selection: Zhengguang 1, Zhengguang 2, GB20, GV14, LI4.
  * plum-blossom needle manipulation methods: After the skin has been wiped with 75 % alcohol, plum-blossom needles will be tapped perpendicularly on the skin at the selected acupoints with wrist force and then lifted immediately. Each point will be tapped repeatedly for 20 to 50 times and both sides of cervical vertebra and temporal region, Suprao-infraorbital margin will be tapped repeatedly. Acupuncturists should tap the points gently to make patients feel only a little pain and stop when the skin gets flushed but is not bleeding.
  Other Names: Double head dermal needles (HWATO, China)
Drug: Tropicamide Eye Drops — Instill one drop in both eyes every night before bed.
  Other Names: 6ml:30mg(0.5%)（FREDA, China）

SUMMARY:
The purpose of this study is to determine whether plum-blossom needle is effective in the treatment of juvenile myopia and compare the efficacy with Tropicamide Eye Drops.

DETAILED DESCRIPTION:
Plum-blossom needle is a historical treatment technology of Traditional Chinese Medicine, and has been applied to ophthalmic diseases, such as myopia and glaucoma, for nearly one hundred years.

ELIGIBILITY:
Inclusion Criteria:

* The result of retinoscopy is myopic refractive error, near visual acuity and other visual functions must be normal
* Distance visual acuity can be corrected to normal using negative spherical or cylindrical lenses
* Myopia diopter spherical lenses must be ≤-3.00 D which measured under cycloplegia
* Subjects must be between 8 and 20 years of age

Exclusion Criteria:

* Diopter spherical lenses be >-3.00 D , or uncorrected distance visual acuity <0.1, or pathologic myopia with eye complications
* Diopter spherical lense ≥1.50 D or cylindrical lenses ≥1.00 D, as measured under cycloplegia
* The affected eyes have other diseases which affect the determination of acupuncture efficacy
* Subjects with serious systemic diseases, such as cerebrovascular, liver, kidney, hematopoietic system, and psychiatric diseases
* Longterm use of other related drugs or treatments, which have not been terminated
* Parents or subjects refuse to participate this trial
* Participating other ongoing clinical trials

Ages: 8 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 98 (Estimated)
Dates: Start 2016-12; Primary Completion 2018-01 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Changes of vision acuity | Every 30 days for 150 days
  International Standard Visual Acuity Chart
Changes of cycloplegic refractive errors | Every 30 days for 150 days
  Measured using subjective refraction

SECONDARY OUTCOMES:
Changes of accommodation responses | Every 30 days for 150 days
Changes of accommodation facility | Every 30 days for 150 days
Changes of ciliary body thickness | Every 30 days for 150 days
Changes of axial length | Every 30 days for 150 days

CONTACTS AND LOCATIONS:
Overall Officials: Yuanbo Liang, Doctor, Study Director — Clinical&Epidemiological Eye Research Center
Locations (1):
- School of Ophthalmology and Optometry, Eye Hospital, Wenzhou Medical University, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided
The IPD sharing plan is undecided yet.

REFERENCES:
- [Derived] Chen L, Liang Y, Xu M, Zheng J, Yu H, Tang L. Effect of plum-blossom needling versus tropicamide eye drops on adolescent myopia: protocol for a randomized crossover trial. J Tradit Chin Med. 2020 Apr;40(2):333-339. PMID 32242400